CLINICAL TRIAL: NCT00115557
Title: Delivery of Preventive Services in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: James Mold, MD, MPH, University of Oklahoma HSC Department of Family and Preventive Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21HS014850 (AHRQ)
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2007-09

CONDITIONS: Preventive Services; Immunizations; Screening
Keywords: translational research; prevention; primary care; practice-based research network

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Performance feedback, academic detailing, practice facilitation, IT support
  Interventions: Other: Practice intervention
- 2 (Active Comparator): Performance feedback only
  Interventions: Other: Practice intervention 2

INTERVENTIONS:
Other: Practice intervention — Performance feedback, academic detailing, practice facilitation, IT support
  Arms: 1
Other: Practice intervention 2 — Performance feedback only.
  Arms: 2

SUMMARY:
The major goal of this project is to determine the effectiveness of a multi-component intervention designed to help primary care practices implement three office system strategies known to increase delivery of immunizations and other preventive services. This two-year study will contribute to our understanding of multi-component translational interventions in primary care, and particularly within practice-based research networks.

DETAILED DESCRIPTION:
The multi-component translational intervention that we plan to test includes medical record audits with feedback and benchmarking, academic detailing by an opinion leader including information from literature review plus the advice of local exemplars, a practice facilitator, who will work with the practices over a six-month period, and an IT application that provides decision-support, prompts, and reminders to office staff and patients.

The proposed project will be a randomized controlled trial of a multi-component strategy designed to facilitate the incorporation into primary care practices of three office management components known to increase preventive service delivery rates: 1) nurse standing orders; 2) special immunization/ preventive services "clinics;" and 3) recall and reminder systems. Twenty-four practices, all members of a primary care practice-based research network, will be enrolled and randomized to receive the complete intervention or performance feedback with benchmarking only. The primary outcomes will be number of management components implemented. Characteristics of clinicians and practices that are associated with greater or lesser success in implementing the three strategies and barriers encountered will also be examined, and we will measure and compare rates of selected immunizations and preventive services delivered.

The specific aims for this project are to:

1. Determine the effectiveness of a multi-component translational intervention on adoption of three strategies known to increase delivery of preventive services: nurse standing orders, a reminder/recall system (preferably PSRS), and special immunization and/or preventive services clinics. The intervention will include: a) performance feedback and benchmarking; b) training of clinicians and office staff in principles of effective preventive services (enhanced academic detailing by a physician opinion leader); c) practice enhancement assistants to facilitate office system changes; and d) an IT application that provides prompts and reminders to office staff, clinicians, and patients.
2. Document contextual factors and barriers to the adoption of the three strategies and their impact on the intervention.
3. Measure the impact of the intervention on rates of delivery of the following preventive services: DtaP#4, MMR#1, and HepB#3 in 2-3 year olds, and pneumococcal immunization, colorectal cancer screening, and mammography in adults 50 - 75 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Primary care physician
* Member of the Oklahoma Physicians Resource/Research Network
* Computer with internet connection
* More than 30 patients seen per week
* Provides care to 2-3 year-olds and/or 50-75 year olds

Exclusion Criteria:

* Does not provide preventive services
* Inclusion of more than two of the preventive service delivery strategies at baseline
* Involved in another network project
* Unwilling to work with an external practice facilitator
* IRB used by the practice will not allow records audits without individual patient consent

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-10; Primary Completion 2006-05 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Implementation of one or more of three evidence-based strategies | 6 months

SECONDARY OUTCOMES:
Rates of delivery of selected preventive services | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James W Mold, MD, MPH, Principal Investigator — University of Oklahoma
Locations (1):
- OKPRN, Oklahoma City, Oklahoma, United States